CLINICAL TRIAL: NCT02384733
Title: The Skagen Trial 1, Moderately Hypofractionated Loco-regional Adjuvant Radiation Therapy of Early Breast Cancer Combined With a Simultaneous Integrated Boost: a Randomised Clinically Controlled Trial
Brief Title: Hypofractionated Loco-regional Adjuvant Radiation Therapy of Breast Cancer Combined With a Simultaneous Integrated Boost
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Breast Cancer Cooperative Group (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Birgitte Offersen, MD, professor, ph.d., Danish Breast Cancer Cooperative Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The Skagen Trial 1
Record Dates: First submitted 2015-02-19; First posted 2015-03-10 (Estimated); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Lymphedema; Fibrosis
Keywords: Radiation induced morbidity, recurrence
MeSH Terms: conditions — Lymphedema; Fibrosis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypofractionated loco-regional RT (Experimental): 40 Gy / 15 fractions, 2.67 Gy per fraction, 5 fractions weekly
  Interventions: Radiation: Loco-regional RT
- Normofractionated loco-regional RT (Active Comparator): 50 Gy / 25 fractions, 2.00 Gy per fraction, 5 fractions weekly
  Interventions: Radiation: Loco-regional RT

INTERVENTIONS:
Radiation: Loco-regional RT

SUMMARY:
The purpose of the study is to investigate the difference in late radiation morbidity between hypofractionated and normofractionated loco-regional breast irradiation irrespective of mastectomy or lumpectomy. In patients who a candidates for a boost, the boost will be provided as a simultaneous integrated boost.

DETAILED DESCRIPTION:
The randomization is between 50 Gy / 25 fractions and 40 Gy/15 fractions, 5 fractions weekly. In patients treated with boost 2 dose levels are accepted: 16 Gy/8 fractions and 10 Gy/5 fractions. These boost treatments will be provided as simultaneous integrated boost, where the overall treatment time in general is shortened 5 days. Thus the dose levels for boost patients are:

63 Gy / 51.52 Gy / 28 fractions, 57 Gy / 50 Gy / 25 fractions, 52.2 Gy / 42.3 Gy / 18 fractions, and 45.75 Gy / 40 Gy / 15 fractions.

The primary endpoint is arm lymphedema 3 years after radiation therapy, but other late radiation morbidities will also be evaluated along with recurrence and sites of recurrence. Follow up of morbidity will continue for 10 years.

The hypothesis is that women operated for early breast cancer with indication for loco-regional radiation therapy can be offered moderately hypofractionated therapy without developing more late radiation induced morbidity compared to normofractionated radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

Operated for early node-positive breast cancer with indication for loco-regional breast radiotherapy

Exclusion Criteria:

Previous radiotherapy to chest wall, pregnant/lactating, comorbidity which may hinder 10 years follow up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2963 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2032-07-01 (Estimated)

PRIMARY OUTCOMES:
Development of ipsilateral arm lymphedema | 3 years
  >=10% increased arm circumference compared to the other arm defines edema

SECONDARY OUTCOMES:
Fibrosis grade 2-3 | 3 years
  Breast or chest wall induration
Arm range of motion | 3 years
  Impaired shoulder movement is present when >20 degrees difference between arms at flexion and/or abduction
Development of dyspigmentation | 3 years
  Grade 2 or worse dyspigmentation compared to baseline
Recurrence | 10 years
  Any recurrence location and time to event
Development of pain in the irradiated area | 3 years
  Pain in the irradiated area measured on visual analog scale compared to baseline
Change in sensibility | 3 years
  Change in sensibility in the irradiated area compared to baseline measured as yes/no
Development of edema on breast / chest wall | 3 years
  Grade 2 or worse edema
Development of telangiectasia in irradiated area | 3 years
  Grade 2 or worse telangiectasia

CONTACTS AND LOCATIONS:
Overall Officials: Lars Stenbygaard, MD, Study Chair — Aalborg University Hospital; Troels Bechmann, MD,PhD, Study Chair — Vejle Hospital; Mette Nielsen, MD, Study Chair — Odense University Hospital; Birgitte Offersen, MD, Principal Investigator — Aarhus University Hospital; Hanne Nielsen, MD, Study Chair — Aarhus University Hospital; Claus Kamby, MD, Study Chair — Rigshospitalet, Denmark; Sami Al-Rawi, MD, Study Chair — Naestved Hospital; Mechthild Krause, MD, Study Chair — Technische Universität Dresden Klinik und Poliklinik für Strahlentherapie und Radioonkologie; Andreas Schreiber, MD, Study Chair — Praxis für Strahlentherapie, Dresden; Ingvil Mjaaland, MD, Study Chair — Stavanger Hospital; Tanja Marinko, MD, Study Chair — Institute of Oncology Ljubljana; Carine Kirkove, MD, Study Chair — Radiotherapy Department Université Catholique de Louvain, Cliniques Universitaires St-Luc, Brussels; Egil Blix, MD, Study Chair — University Hospital of North Norway, Tromsoe; Unn-Miriam Kasti, Study Chair — Kristiansand Hospital, Norway
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark